CLINICAL TRIAL: NCT07193277
Title: Safety and Efficacy of Butylphthalide Soft Capsules for Cognitive Impairment Comorbid With Focal Epilepsy in Elderly Patients: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Butylphthalide for Cognitive Impairment in Elderly Patients With Focal Epilepsy
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Collaborators: Taizhou Hospital (Other); Lishui Country People's Hospital (Other); Affiliated Yueqing Hospital of Wenzhou Medical University (Other); The Third Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KY2025-330
Record Dates: First submitted 2025-09-10; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Focal Epilepsy; Cognitive Impairment
Keywords: Butylphthalide; Focal Epilepsy; Cognitive Impairment; Elderly; MoCA; Neuroprotection; Randomized Controlled Trial; Double-blind; Placebo-controlled; Multicenter
MeSH Terms: conditions — Epilepsies, Partial; Cognitive Dysfunction | interventions — 3-n-butylphthalide

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1 ratio to receive either butylphthalide soft capsules or matching placebo for 48 weeks. Both groups will continue their stable anti-seizure medication regimen throughout the study period.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind design where participants, care providers, investigators, and outcomes assessors are masked to treatment assignment. Emergency unblinding procedures are available when medically necessary.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Butylphthalide Group (Experimental): Participants receive butylphthalide soft capsules 0.2g (two 0.1g capsules) orally three times daily before meals for 48 weeks, while continuing their stable anti-seizure medication regimen.
  Interventions: Drug: Butylphthalide
- Placebo Group (Placebo Comparator): Participants receive matching placebo capsules orally three times daily before meals for 48 weeks, while continuing their stable anti-seizure medication regimen. Placebo capsules are identical in appearance, weight, and odor to butylphthalide capsules.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Butylphthalide — Butylphthalide soft capsules (0.1g per capsule) manufactured by CSPC NBP Pharmaceutical Co., Ltd. Participants take 2 capsules (0.2g total) orally three times daily, 15-30 minutes before meals, for 48 weeks. This represents off-label use for cognitive impairment comorbid with epilepsy, as the drug is currently approved in China only for acute ischemic stroke treatment.
  Other Names: DL-3-n-butylphthalide; NBP
  Arms: Butylphthalide Group
Drug: Placebo — Matching placebo capsules identical in appearance, weight, and odor to butylphthalide soft capsules, manufactured by the same company following GMP standards. Participants take 2 capsules orally three times daily, 15-30 minutes before meals, for 48 weeks. Placebo contains starch and appropriate excipients.
  Arms: Placebo Group

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled trial evaluating the safety and efficacy of butylphthalide soft capsules for treating cognitive impairment in elderly patients with focal epilepsy.

Study Population: 220 elderly patients (60-85 years) with focal epilepsy and mild to moderate cognitive impairment (Montreal Cognitive Assessment score 18-25).

Intervention: Participants will be randomly assigned 1:1 to receive either butylphthalide soft capsules (0.2g three times daily) or matching placebo for 48 weeks, while continuing their stable anti-seizure medication regimen.

Primary Outcome: Change in Montreal Cognitive Assessment (MoCA) total score from baseline to 48 weeks.

Secondary Outcomes: Changes in neuropsychological tests (Trail Making Test, Digit Span, Rey Auditory Verbal Learning Test), seizure control measures, functional status (Activities of Daily Living, Quality of Life in Epilepsy), and exploratory neurobiological markers.

This study addresses an important unmet medical need, as current epilepsy treatments focus primarily on seizure control but lack effective interventions for epilepsy-associated cognitive impairment. Butylphthalide, a neuroprotective agent approved for acute ischemic stroke in China, has shown promise in other cognitive disorders and may benefit this patient population through its multiple neuroprotective mechanisms.

DETAILED DESCRIPTION:
Background and Rationale:

Epilepsy affects approximately 9 million people in China, with focal epilepsy comprising 60-70% of adult cases. Cognitive impairment occurs in 40-60% of elderly patients with focal epilepsy, significantly impacting quality of life and daily functioning. Current anti-seizure medications effectively control seizures in ~70% of patients but provide limited benefit for cognitive symptoms, and some may even worsen cognitive function.

Butylphthalide (DL-3-n-butylphthalide) is a multi-target neuroprotective compound originally derived from celery seeds, approved in China for acute ischemic stroke treatment. Its mechanisms include improving cerebral microcirculation, protecting mitochondrial function, reducing oxidative stress, anti-inflammatory effects, and anti-apoptotic properties. Previous studies have demonstrated efficacy in vascular cognitive impairment and mild cognitive impairment, but its effects in epilepsy-associated cognitive dysfunction remain unexplored.

Study Design:

This investigator-initiated, multicenter, randomized, double-blind, placebo-controlled trial will enroll 220 participants across 5 centers in China. The study represents off-label use of butylphthalide for cognitive impairment comorbid with epilepsy.

Participants will undergo comprehensive cognitive assessment including MoCA, Trail Making Tests A/B, Digit Span (forward/backward), Rey Auditory Verbal Learning Test, Activities of Daily Living scale, and Quality of Life in Epilepsy inventory. Exploratory endpoints include functional near-infrared spectroscopy, electroencephalography parameters, and serum biomarkers (BDNF, NGF, NSE, S100β, inflammatory markers).

The 48-week treatment period reflects the chronic nature of cognitive impairment and allows adequate time to detect clinically meaningful changes. Safety monitoring includes regular laboratory assessments, vital signs, and adverse event reporting. A 24-hour emergency contact system ensures participant safety.

Statistical Considerations:

Sample size calculation is based on a minimal clinically important difference of 2.5 points on the MoCA scale, with 80% power and 20% dropout rate. Primary analysis uses ANCOVA comparing 48-week MoCA change scores between groups, adjusting for baseline values and study center. Mixed-effects models will analyze repeated measures for secondary endpoints.

This study may provide evidence for a novel therapeutic approach to epilepsy-associated cognitive impairment, potentially expanding treatment options for this underserved patient population.

ELIGIBILITY:
Inclusion Criteria:

* Age 60-85 years (inclusive)
* Diagnosed with focal epilepsy according to ILAE 2025 latest classification standards, with disease duration ≥2 years
* Currently receiving stable anti-seizure medication (ASM) treatment for ≥3 months, with good seizure control (monthly seizure frequency ≤4 times in the past 3 months)
* Cognitive impairment: Montreal Cognitive Assessment (MoCA) score 18-25 points (inclusive)
* Basic Chinese language comprehension and expression ability, able to cooperate with neuropsychological testing
* Voluntary participation and signed informed consent

Exclusion Criteria:

* Diagnosed with various types of dementia (including Alzheimer's disease, vascular dementia, etc.)
* Clear history of stroke with corresponding lesions on neuroimaging, or severe white matter lesions on brain MRI
* Other neurological diseases that may cause cognitive impairment (traumatic brain injury, encephalitis, hydrocephalus, etc.)
* Systemic diseases that may cause cognitive impairment (severe cardiac, hepatic, renal dysfunction, endocrine diseases, etc.)
* Current severe depression or other psychiatric diseases affecting cognitive assessment
* History of alcohol dependence, drug abuse, or other substance use affecting cognitive function
* Allergy to butylphthalide or its excipients
* Participation in other drug clinical trials within 30 days
* Other conditions deemed inappropriate for participation by investigators

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Montreal Cognitive Assessment (MoCA) Total Score from Baseline to 48 Weeks | Baseline and 48 weeks
  The Montreal Cognitive Assessment (MoCA) is a validated cognitive screening tool that evaluates multiple cognitive domains including visuospatial/executive function, naming, memory, attention, language, abstraction, delayed recall, and orientation. The total score ranges from 0 to 30 points, with higher scores indicating better cognitive function. The primary outcome is the change in MoCA total score from baseline to 48 weeks, calculated as: (MoCA score at 48 weeks) - (MoCA score at baseline). A positive change indicates cognitive improvement, while a negative change indicates cognitive decline.

SECONDARY OUTCOMES:
Trail Making Test Part A (TMT-A) Completion Time Changes | Baseline, 12 weeks, 24 weeks, 36 weeks, and 48 weeks
  Trail Making Test Part A (TMT-A) assesses visual scanning speed and psychomotor speed. Participants connect numbered circles in ascending order (1-2-3-4-5...-25). Completion time is measured in seconds, with typical ranges from 15-300 seconds depending on age and education. Lower completion times indicate better performance. The outcome is calculated as: (TMT-A time at assessment point) - (TMT-A time at baseline). A negative change indicates improvement.
Trail Making Test Part B (TMT-B) Completion Time Changes | Baseline, 12 weeks, 24 weeks, 36 weeks, and 48 weeks
  Trail Making Test Part B (TMT-B) assesses executive function including cognitive flexibility and attention switching. Participants alternate between numbers and letters (1-A-2-B-3-C...). Completion time is measured in seconds, with typical ranges from 30-600 seconds depending on age and education. Lower completion times indicate better performance. The outcome is calculated as: (TMT-B time at assessment point) - (TMT-B time at baseline). A negative change indicates improvement.
Digit Span Forward Test Score Changes | Baseline, 12 weeks, 24 weeks, 36 weeks, and 48 weeks
  Digit Span Forward Test assesses attention and short-term memory capacity. Participants repeat number sequences in the same order as presented. Scores range from 0 to 9 points, with higher scores indicating better attention and short-term memory performance. The outcome is calculated as: (Digit Span Forward score at assessment point) - (Digit Span Forward score at baseline). A positive change indicates improvement.
Digit Span Backward Test Score Changes | Baseline, 12 weeks, 24 weeks, 36 weeks, and 48 weeks
  Digit Span Backward Test assesses working memory and mental manipulation abilities. Participants repeat number sequences in reverse order. Scores range from 0 to 8 points, with higher scores indicating better working memory performance. The outcome is calculated as: (Digit Span Backward score at assessment point) - (Digit Span Backward score at baseline). A positive change indicates improvement.
Rey Auditory Verbal Learning Test (RAVLT) Immediate Recall Score Changes | Baseline, 12 weeks, 24 weeks, 36 weeks, and 48 weeks
  Rey Auditory Verbal Learning Test (RAVLT) Immediate Recall assesses verbal learning and immediate memory capacity. Participants recall a 15-word list immediately after the fifth presentation. Scores range from 0 to 15 words correctly recalled, with higher scores indicating better immediate verbal memory performance. The outcome is calculated as: (RAVLT immediate recall score at assessment point) - (RAVLT immediate recall score at baseline). A positive change indicates improvement.
Rey Auditory Verbal Learning Test (RAVLT) Delayed Recall Score Changes | Baseline, 12 weeks, 24 weeks, 36 weeks, and 48 weeks
  Rey Auditory Verbal Learning Test (RAVLT) Delayed Recall assesses long-term verbal memory retention. Participants recall the 15-word list after a 30-minute delay. Scores range from 0 to 15 words correctly recalled, with higher scores indicating better long-term verbal memory performance. The outcome is calculated as: (RAVLT delayed recall score at assessment point) - (RAVLT delayed recall score at baseline). A positive change indicates improvement.
Average Monthly Seizure Frequency Percentage Change | Baseline, 12 weeks, 24 weeks, 36 weeks, and 48
  Percentage change in average monthly seizure frequency from baseline to each assessment timepoint. Seizure frequency is recorded daily through seizure diary maintained by patients and caregivers, verified during clinical visits. The outcome is calculated as: [(Average monthly frequency at assessment point) - (Average monthly frequency at baseline)] / (Average monthly frequency at baseline) × 100%. A negative percentage indicates reduction in seizure frequency (improvement).
Proportion of Participants with ≥50% Reduction in Seizure Frequency | Baseline and 48 weeks
  Percentage of participants achieving at least 50% reduction in average monthly seizure frequency compared to baseline. Response is defined as: (Baseline monthly frequency - Average monthly frequency during weeks 45-48) / Baseline monthly frequency ≥ 50%. Seizure data collected through daily seizure diary and verified by caregivers.
Activities of Daily Living (ADL) Scale Score Changes | Baseline, 12 weeks, 24 weeks, 36 weeks, and 48 weeks
  Activities of Daily Living (ADL) Scale is a 14-item assessment tool that evaluates both basic activities of daily living (BADL) including feeding, bathing, grooming, dressing, bowel control, and bladder control, and instrumental activities of daily living (IADL) including using telephone, shopping, food preparation, housekeeping, laundry, transportation, medication responsibility, and financial management. Each item is scored from 1 to 4 points, with total scores ranging from 14 to 56 points. Higher scores indicate greater functional impairment (worse outcome). The outcome is calculated as: (ADL score at assessment point) - (ADL score at baseline). A negative change indicates functional improvement.
Quality of Life in Epilepsy Inventory-31-Patient weighted (QOLIE-31-P) Score Changes | Baseline, 12 weeks, 24 weeks, 36 weeks, and 48 weeks
  Quality of Life in Epilepsy Inventory-31-Patient weighted (QOLIE-31-P) evaluates epilepsy-specific quality of life across 7 domains: seizure worry, overall quality of life, emotional well-being, energy/fatigue, cognitive functioning, medication effects, and social function. Total scores range from 0 to 100 points, with higher scores indicating better quality of life. The outcome is calculated as: (QOLIE-31-P score at assessment point) - (QOLIE-31-P score at baseline). A positive change indicates improvement.
Number of Participants with Treatment-Related Adverse Events as Assessed by Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0) | 12 weeks, 24 weeks, 36 weeks, and 48 weeks
  Safety and tolerability assessed by incidence of treatment-related adverse events classified and graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. All adverse events will be recorded and their relationship to study drug will be assessed by investigators as unrelated, unlikely, possible, probable, or definite.
Number of Participants with Serious Adverse Events | 12 weeks, 24 weeks, 36 weeks, and 48 weeks
  Incidence of serious adverse events (SAEs) defined according to International Conference on Harmonisation (ICH) guidelines as events that result in death, are life-threatening, require inpatient hospitalization or prolongation of existing hospitalization, result in persistent or significant disability/incapacity, are congenital anomaly/birth defect, or are medically important events.
Number of Participants with Clinically Significant Hepatic Function Abnormalities | 24 weeks and 48 weeks
  Incidence of clinically significant hepatic function abnormalities defined as alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels greater than 2 times the upper limit of normal (ULN), or total bilirubin greater than 1.5 times ULN as measured by standard laboratory methods.
Number of Participants with Clinically Significant Renal Function Abnormalities | 24 weeks and 48 weeks
  Incidence of clinically significant renal function abnormalities defined as serum creatinine levels greater than 1.5 times the upper limit of normal (ULN) or estimated glomerular filtration rate (eGFR) decrease by ≥25% from baseline as measured by standard laboratory methods.
Number of Participants with Clinically Significant Hematological Abnormalities | 24 weeks and 48 weeks
  Incidence of clinically significant hematological abnormalities including hemoglobin decrease to less than 11 g/dL, white blood cell count less than 3,000/μL or greater than 11,000/μL, or platelet count less than 100,000/μL or greater than 450,000/μL as measured by standard hematology laboratory methods.

CONTACTS AND LOCATIONS:
Overall Officials: Huiqin Xu, MD, Principal Investigator — Department of Neurology, First Affiliated Hospital of Wenzhou Medical University
Locations (1):
- First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided
The data sharing plan is currently under consideration and will be determined in consultation with all participating centers, institutional review boards, and relevant regulatory authorities. Factors being evaluated include compliance with Chinese data protection regulations, patient consent provisions, and journal publication policies. A final decision on individual participant data sharing will be made prior to study completion and updated in this registration record.